CLINICAL TRIAL: NCT00722540
Title: Dose Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NCC126-0083 in Healthy Male Japanese Subjects.
Brief Title: Dose Study in Healthy Japanese Males Investigating Safety, Pharmacokinetics and Pharmacodynamics of NNC126-0083
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8630-1958; 2008-001578-33 (EudraCT Number)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Healthy
MeSH Terms: interventions — NNC126-0083

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- B (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- C (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- D (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo
- E (Experimental)
  Interventions: Drug: NNC126-0083; Drug: placebo

INTERVENTIONS:
Drug: NNC126-0083 — Dose level 1; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Arms: A
Drug: NNC126-0083 — Dose level 2; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Arms: B
Drug: NNC126-0083 — Dose level 3; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Arms: C
Drug: NNC126-0083 — Dose level 3 repeated; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: D
Drug: placebo — Dose level 1; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: A
Drug: placebo — Dose level 2; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: B
Drug: placebo — Dose level 3; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: C
Drug: placebo — Dose level 3 repeated; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: D
Drug: NNC126-0083 — Dose level 4; (6 subjects active, 2 subjects placebo); s.c. injection once weekly for 3 weeks
  Arms: E
Drug: placebo — Dose level 4; NNC126-0083 placebo for s.c. injection once weekly for 3 weeks
  Arms: E

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of a NNC126-0083 in healthy male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects with Japanese passport and Japanese born parents
* Body Mass Index (BMI, kg/m2) between 18.0 and 27.0, both inclusive
* Subjects must be in good health according to age

Exclusion Criteria:

* A history or presence of cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major diseases
* History of any illnesses or disease that, in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the trial product to the subject
* Any clinically significant abnormal haematology, biochemistry or urinalysis screening tests, as judged by the Investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events, local tolerability, physical examination) | 0 to 10 days after third dosing, (day 15-25 after first dose)

SECONDARY OUTCOMES:
Cmax, maximum concentration of IGF-I | 7 days after first dosing and 10 days after the third dosing (day 1-25 after first dose)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Rasmussen MH, Jensen L, Anderson TW, Klitgaard T, Madsen J. Multiple doses of pegylated long-acting growth hormone are well tolerated in healthy male volunteers and possess a potential once-weekly treatment profile. Clin Endocrinol (Oxf). 2010 Dec;73(6):769-76. doi: 10.1111/j.1365-2265.2010.03863.x. PMID 20718773
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com